CLINICAL TRIAL: NCT00917540
Title: Prospective Collection of Biological Data of Prognostic Relevance in Patients
Brief Title: Prospective Collection of Biological Data of Prognostic Relevance in Patients With B-Cell Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Sponsor
Other Study IDs: O-CLL1
Record Dates: First submitted 2009-05-08; First posted 2009-06-10 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Lymphocytic Leukemia Stage A(0); Chronic Lymphocytic Leukemia Stage A(I); Chronic Lymphocytic Leukemia Stage A(II)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the present study is to develop a biological prognostic index in patients with Binet stage A Chronic Lymphocytic Leukemia (CLL) who do not necessitate therapy according to NCI guidelines and to prospectively validate the proposed score system based on the absence/presence of 1, 2 or 3 unfavorable prognostic markers such as cluster of differentiation 38 (CD38) expression, Zap-70 expression and immunoglobulin heavy chain variable region (IgVH) configuration.

DETAILED DESCRIPTION:
Clinical data including information on disease localization and laboratory parameters will be collected at study entry, during follow up and at disease progression (or after 36 months after registration) Biological markers will be evaluated at centralized laboratory, at study entry and at time of disease progression (or after 24 months of follow-up for non progressed patients) Using the scoring system, patients can be separated into 3 risk groups: low-risk (score 0), intermediate-risk (score 1) and high-risk (score 2-3), with significantly different clinical courses.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of B-CLL by NCI criteria, performed by local haematologist. (Diagnosis will be confirmed by the biological review committee according to flow cytometry analysis (positive clusters of differentiation antigen 5 (CD5), 19 (CD19),23 (CD23)).
* Age > 18 years and < 70 years.
* Eastern Cooperative Oncology Group (ECOG)<=2.
* Binet stage A.
* Diagnosis performed within 12 months before inclusion in the study.
* Patients who do not necessitate therapy by NCI guidelines (watch and wait policy).
* Shipment of peripheral blood sample to centralized laboratory for biological assessment.
* Clinical data including baseline information on disease localization and laboratory parameters at staging and assurance of follow up updating for at least 3 years are requested.
* Written informed consent.

Exclusion Criteria:

* Patients with CLL whose diagnosis exceed 12 months before registration.
* Patients with leukemic phase of lymphoproliferative disorders of B origin CD5- and/or CD23- according to flow cytometry analysis.
* Clinical Binet stage B or C.
* Patients who necessitate therapy according to NCI guide-lines (no watch and wait policy).
* Age > 70 years.
* Without a written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated Binet stage A B-CLL patients, who do not necessitate therapy according to NCI guidelines
Sampling Method: Non-Probability Sample
Enrollment: 495 (Estimated)
Dates: Start 2007-02; Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Prospective validation of the prognostic potential of a score system based on the presence/absence of three risk factors (VH mutational status, Zap-70 and CD38 expression) on Progression Free Survival (PFS ). | 6 months

SECONDARY OUTCOMES:
Quality of Life | 6 months
Time to Treatment | 6 months
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Morabito, MD, Study Chair — GISL; Manlio Ferrarini, MD, Study Chair — GISL
Locations (1):
- GISL Trial Office, Modena, Italy

REFERENCES:
- [Derived] Matis S, Grazia Recchia A, Colombo M, Cardillo M, Fabbi M, Todoerti K, Bossio S, Fabris S, Cancila V, Massara R, Reverberi D, Emionite L, Cilli M, Cerruti G, Salvi S, Bet P, Pigozzi S, Fiocca R, Ibatici A, Angelucci E, Gentile M, Monti P, Menichini P, Fronza G, Torricelli F, Ciarrocchi A, Neri A, Fais F, Tripodo C, Morabito F, Ferrarini M, Cutrona G. MiR-146b-5p regulates IL-23 receptor complex expression in chronic lymphocytic leukemia cells. Blood Adv. 2022 Oct 25;6(20):5593-5612. doi: 10.1182/bloodadvances.2021005726. PMID 35819446
- [Derived] Morabito F, Tripepi G, Vigna E, Bossio S, D'Arrigo G, Martino EA, Storino F, Recchia AG, Fronza G, Di Raimondo F, Colombo M, Fais F, Neri A, Cutrona G, Ferrarini M, Gentile M. Validation of the Alternative International Prognostic Score-E (AIPS-E): Analysis of Binet stage A chronic lymphocytic leukemia patients enrolled into the O-CLL1-GISL protocol. Eur J Haematol. 2021 Jun;106(6):831-835. doi: 10.1111/ejh.13614. Epub 2021 Apr 7. PMID 33662164
- [Derived] Kreuzberger N, Damen JA, Trivella M, Estcourt LJ, Aldin A, Umlauff L, Vazquez-Montes MD, Wolff R, Moons KG, Monsef I, Foroutan F, Kreuzer KA, Skoetz N. Prognostic models for newly-diagnosed chronic lymphocytic leukaemia in adults: a systematic review and meta-analysis. Cochrane Database Syst Rev. 2020 Jul 31;7(7):CD012022. doi: 10.1002/14651858.CD012022.pub2. PMID 32735048
- [Derived] Morabito F, Cutrona G, Mosca L, D'Anca M, Matis S, Gentile M, Vigna E, Colombo M, Recchia AG, Bossio S, De Stefano L, Maura F, Manzoni M, Ilariucci F, Consoli U, Vincelli I, Musolino C, Cortelezzi A, Molica S, Ferrarini M, Neri A. Surrogate molecular markers for IGHV mutational status in chronic lymphocytic leukemia for predicting time to first treatment. Leuk Res. 2015 Aug;39(8):840-5. doi: 10.1016/j.leukres.2015.05.005. Epub 2015 May 19. PMID 26038121
- [Derived] Maura F, Mosca L, Fabris S, Cutrona G, Matis S, Lionetti M, Agnelli L, Barbieri M, D'Anca M, Manzoni M, Colombo M, Massucco C, Reverberi D, Gentile M, Recchia AG, Bossio S, Ilariucci F, Musolino C, Di Raimondo F, Cortelezzi A, Morabito F, Ferrarini M, Neri A. Insulin growth factor 1 receptor expression is associated with NOTCH1 mutation, trisomy 12 and aggressive clinical course in chronic lymphocytic leukaemia. PLoS One. 2015 Mar 18;10(3):e0118801. doi: 10.1371/journal.pone.0118801. eCollection 2015. PMID 25786252